CLINICAL TRIAL: NCT05945004
Title: Using Natural Language Processing Models for Writing Preoperative Visit Sheets: a Preliminary Study Comparing ChatGPT and Clinicians
Brief Title: ChatGPT v.s. Human in Writing a Preoperative Visit Sheet
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Boston Intelligent Medical Research Center, Shenzhen United Scheme Technology Co., Ltd. (Industry)
Collaborators: Tsinghua University (Other)
Responsible Party: Sponsor
Other Study IDs: US2023002
Record Dates: First submitted 2023-06-30; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Preoperative Care
MeSH Terms: interventions — Nurse Clinicians

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experiment
  Interventions: Other: ChatGPT-4
- Control
  Interventions: Other: Clinician

INTERVENTIONS:
Other: ChatGPT-4 — Subjects' clinical records will be read by ChatGPT-4 to write preoperative visit sheets.
  Groups: Experiment
Other: Clinician — Subjects' clinical records will be read by clinicians to write preoperative visit sheets.
  Groups: Control

SUMMARY:
The goal of this study is to evaluate the performance of large language models i.e. ChatGPT, in making preoperative visit sheets using clinical records. The main questions it aims to answer are:

* Can large language models read clinical records and make preoperative visit sheets same as physicians?
* Can physicians distinguish preoperative visit sheets made by physicians and models?

Participants' records will be generated using ChatGPT-4, and read by both ChatGPT-4 and physicians to make 2 separate preoperative visit sheets, and form 2 groups, GPT group and physician group respectively.

A group of professionals will compare result of above mentioned 2 groups to see if ChatGPT can afford to write preoperative visit sheets.

ELIGIBILITY:
Inclusion Criteria:

* Any as records are generated using ChatGPT-4.

Exclusion Criteria:

* Any as records are generated using ChatGPT-4.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No restictions are applied to population.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Familiarity to human writing | Each record will be screened for 6 minutes at most and results will be given in 8 minutes after receiving a record.
  Based on professionals' subjective evaluation, familiarity is a binary result indicating weather professionals think the preoperative visit sheet was written by physicians or ChatGPT, where 0 indicates "not written by human" and 1 indicates "written by human".
Satisfaction for clinical use | Each record will be screened for 6 minutes at most and results will be given in 8 minutes after receiving a record.
  A grading score of 1-10 indicating weather the professionals think the preoperative visit sheet is suitable in clinical use.